CLINICAL TRIAL: NCT03209973
Title: A Single Arm, Multicenter, Phase 2 Study of BGB-A317 as Monotherapy in Relapsed or Refractory Classical Hodgkin Lymphoma
Brief Title: A Study of Tislelizumab as Monotherapy in Relapsed or Refractory Classical Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-203; CTR20170119 (Registry Identifier: Center for drug evaluation, CFDA)
Record Dates: First submitted 2017-05-25; First posted 2017-07-06 (Actual); Results first posted 2020-10-12 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab (Experimental): Tislelizumab 200 mg administered intravenously (IV) every-3-weeks (Q3W)
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Administered as specified in the treatment arm
  Other Names: BGB-A317

SUMMARY:
The primary objective of this study was to evaluate the efficacy of tislelizumab assessed by Independent Review Committee (IRC) in participants with relapsed or refractory classical Hodgkin lymphoma (cHL), as measured by Overall Response Rate (ORR) per the Lugano Classification

DETAILED DESCRIPTION:
This was an open-label, single-arm, multi-center Phase 2 study. Response was to be assessed by PET(positron emission tomography) and computed tomography (CT) scan per the Lugano Classification. CT scan with contrast and Positron emission tomography (PET)/CT was used as required by protocol, until progressive disease (PD), new anti-cancer therapy, withdrawal of consent, death, lost to follow-up, or end of study (EOS), whichever occurred first. Total body magnetic resonance imaging (MRI) was allowed if CT with contrast is contraindicated. During treatment with immune checkpoint inhibitor such as with tislelizumab, pseudo-progression may occur due to immune cell infiltration and other mechanisms as manifested by apparent increase of existing tumor masses or appearance of new tumor lesions. Participants were allowed to continue study treatment if there is suspicion of pseudo-progression, provided they are asymptomatic and have radiographic progression only, until a second consecutive CT scan demonstrates PD at which time study treatment was discontinued permanently. Participants were evaluated for Adverse Events (AEs) (all Grades per National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.03 [NCI CTCAE v. 4.03]), serious AEs (SAEs), and any AEs requiring study drug interruption or discontinuation.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed relapsed or refractory cHL (biopsy from diagnosis or at any relapse is acceptable).
2. Participants must have relapsed (disease progression after most recent therapy) or refractory (failure to achieve complete Response (CR) /complete metabolic response [CMR] or partial response (PR) to most recent therapy) cHL and and failed to achieve a response or progressed after auto-SCT or meet the criteria of ineligible for auto-SCT.
3. Participants must have measurable disease defined as ≥ 1 nodal lesion that is > 1.5 cm in the longest diameter, or ≥ 1 extra-nodal lesion (e.g. hepatic nodules) that is > 1 cm in the longest diameter.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Life expectancy ≥ 12 weeks.
6. participants must have adequate organ functions as indicated by the following laboratory values:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, independent of growth factor support within 7 days of first dose.
   2. Platelet ≥ 75 x 109/L, independent of growth factor support or transfusion within 7 days of first dose.
   3. Hemoglobin (Hgb) ≥ 8 g/dL or ≥ 5 mmol/L.
   4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN).
   5. Aspartate aminotransferase (AST)/glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/glutamic-pyruvic transaminase (SGPT) ≤ 2.5 x upper limit of normal (ULN), or ≤ 5X ULN if liver metastases are present.
   6. Serum total bilirubin ≤ 1.5 x ULN (total bilirubin level < 4 x ULN for participants with Gilbert's syndrome).
7. International normalized ratio (INR) ≤ 1.5 x ULN and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless participant is receiving anticoagulant therapy and coagulation parameters (prothrombin time [PT/INR] and aPTT) are within intended therapeutic range of intended use of the anticoagulant at time of Screening. Participants with factor inhibitors prolonging PT or INR may be included after discussion with the medical monitor.
8. Participants must have no evidence of dyspnea at rest and a pulse oximetry of > 92% while breathing room air.
9. Participants must have forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) > 60% by pulmonary function test (PFT); carbon monoxide diffusion capacity (DLCO), FEV1 and FVC all > 50 % predicted value; all PFTs must be obtained within 4 weeks prior to the first dose of tislelizumab.
10. Prior chemotherapy, radiotherapy, immunotherapy or investigational therapy (including Chinese herbal medicine and Chinese patent medicine) used to control cancer including locoregional treatment must have been completed ≥ 4 weeks before the first dose of tislelizumab, and all treatment-related adverse events are stable and have either returned to baseline or Grade 0/1 (except for alopecia and hemoglobin. For hemoglobin, please follow inclusion criteria #8c [hemoglobin]).

Key Exclusion Criteria:

1. Nodular lymphocyte-predominant Hodgkin lymphoma or gray zone lymphoma.
2. Prior allogeneic hematopoietic stem cell transplant.
3. History of severe hypersensitivity reaction to monoclonal antibodies.
4. New York Heart Association (NYHA) class III or IV heart failure, unstable angina, severe uncontrolled ventricular arrhythmia, electrocardiographic evidence of acute ischemia, or myocardial infarction within 6 months of first day of Screening.
5. Prior malignancy within the past 3 years except for curatively treated basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast.
6. Prior therapy targeting PD-1 or PD-L1.
7. Participants with active autoimmune disease or history of autoimmune disease with high risk of recurrence including but not limited to history of immune-related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barrè syndrome, myasthenia gravis, systemic lupus erythematosus (SLE), connective tissue disease, scleroderma, inflammatory bowel disease including Crohn's disease and ulcerative colitis, autoimmune hepatitis, toxic epidermal necrolysis (TEN), or Stevens-Johnson syndrome.

   Note: Participants is permitted to enroll if he/she has vitiligo, eczema, type I diabetes mellitus, endocrine deficiencies including thyroiditis managed with replacement hormone and/or physiologic corticosteroid. Participants with rheumatoid arthritis and/or other arthropathies, Sjögren's syndrome or psoriasis controlled with topical medication, and participants with positive serology such as positive antinuclear antibody (ANA) or anti-thyroid antibody should be evaluated for presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.
8. Conditions requiring systemic treatment with either corticosteroids (> 10 mg daily Prednisone equivalent) or other immunosuppressive medications within 14 days of first dose of tislelizumab.

   Note: Adrenal replacement doses of ≤ 10 mg daily Prednisone are permitted in the absence of active autoimmune disease. Topical, ocular, intra-articular, intra-nasal and inhalational corticosteroid (with minimal systemic absorption), a brief course of corticosteroid for prophylaxis (e.g. contrast dye allergy) or for treatment of non-autoimmune conditions (e.g. delayed-type hypersensitivity reaction caused by contact allergen) are allowed.
9. Has history of interstitial lung disease or non-infectious pneumonitis or has evidence of interstitial lung disease or non infectious pneumonitis currently.
10. QT Interval Corrected by the Fridericia Correction Formula (QTcF)interval > 480 msec, unless secondary to bundle branch block.
11. Serious acute or chronic infection requiring systemic therapy.
12. Known central nervous system (CNS) lymphoma.
13. Underlying medical conditions that, in the Investigator's opinion, will render the administration of study drug hazardous or obscure the interpretation of toxicity or adverse events.
14. Autologous hematopoietic stem cell transplant within 100 days of first dose of tislelizumab.
15. Use of any live vaccine against infectious diseases (e.g. influenza, varicella, etc.) within 4 weeks (28 days) of the first dose of tislelizumab, and any intended use within 60 days after the last dose of tislelizumab.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (12):
- China (12):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chinese Pla General Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Song Y, Gao Q, Zhang H, Fan L, Zhou J, Zou D, Li W, Yang H, Liu T, Wang Q, Lv F, Guo H, Yang L, Elstrom R, Huang J, Novotny W, Wei V, Zhu J. Treatment of relapsed or refractory classical Hodgkin lymphoma with the anti-PD-1, tislelizumab: results of a phase 2, single-arm, multicenter study. Leukemia. 2020 Feb;34(2):533-542. doi: 10.1038/s41375-019-0545-2. Epub 2019 Sep 13. PMID 31520078
- [Derived] Song Y, Gao Q, Zhang H, Fan L, Zhou J, Zou D, Li W, Yang H, Liu T, Wang Q, Lv F, Guo H, Zhao X, Wang D, Zhang P, Wang Y, Wang L, Liu T, Zhang Y, Shen Z, Huang J, Zhu J. Tislelizumab for Relapsed/Refractory Classical Hodgkin Lymphoma: 3-Year Follow-up and Correlative Biomarker Analysis. Clin Cancer Res. 2022 Mar 15;28(6):1147-1156. doi: 10.1158/1078-0432.CCR-21-2023. PMID 34716199
- [Derived] Chen J, Zhang H, Zhu L, Zhao Y, Ding Y, Yuan Y. Tislelizumab for the treatment of classical Hodgkin's lymphoma. Drugs Today (Barc). 2020 Dec;56(12):781-785. doi: 10.1358/dot.2020.56.12.3233362. PMID 33332484

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 participants were enrolled at 11 sites in China. The first participant dose date was on 21 April 2017. The study was completed on 02 November 2020.
Groups:
- Tislelizumab: Tislelizumab 200 mg administered intravenously (IV) every-3-weeks (Q3W) until progressive disease (PD), unacceptable toxicity, death, or study withdrawal by the participant.
Period: Overall Study
Arm/Group | Tislelizumab
Started | 70
Completed Primary Outcome Period | 66
Completed | 0
Not Completed | 70
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 2
Not completed — Death | 8
Not completed — Transferred to Long Term Extension (LTE) study | 32
Not completed — Sponsor Decision | 18
Not completed — Participant Withdrew Due to Higher Risk than Benefit of Treatment | 1
Not completed — Participant Refused to Return to Treatment | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All participants who received any dose of study drug.
Groups:
- Tislelizumab: Tislelizumab 200 mg administered IV Q3W until PD, unacceptable toxicity, death, or study withdrawal by the participant.
Arm/Group | Tislelizumab
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (12.73)
Age, Customized [Count of Participants; unit: Participants]
  <65 | 66
  ≥ 65 and < 75 years | 4
  ≥ 75 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 70
Region of Enrollment [Count of Participants; unit: Participants]
  China | 70

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the proportion of participants who achieve a best response of Complete Response (CR) or Partial Response (PR), as assessed by Independent Review committee (IRC) per the Lugano Classification
Time Frame: From the date of first dose Up to approximately 3 year and 7 months
Population: Modified Safety Analysis Set: All participants in the safety analysis set who had confirmed classical Hodgkin lymphoma.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 70
Percentage of Participants | 87.1 [77.0 to 93.9]
Statistical Analysis 1: Comparison: Tislelizumab; Test type: Other; p < 0.0001, Exact Binomial Test — 1-sided p-value was based on exact test of BGB-A317 versus historical rate of 0.35; Comparison with historical control values

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from the first dose of tislelizumab to the date of Progressive Disease (PD) or death, whichever occurs first, assessed by IRC per the Lugano Classification
Time Frame: From the date of first dose until end of study (Up to approximately 3 years and 7 months)
Population: Modified Safety Analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab
Number analyzed (Participants) | 70
Months | 31.5 [16.53 to NA] — NA = upper limit of confidence interval not estimable due to insufficient event number greater than median value

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the date that response criteria are first met to the date that PD is objectively documented or death, whichever occurs first, assessed by IRC per the Lugano Classification
Time Frame: From the date of first dose until end of study (Up to approximately 3 years and 7 months)
Population: Modified Safety Analysis set; Participants with available data were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab
Number analyzed (Participants) | 61
Months | 31.3 [20.73 to NA] — NA = upper limit of confidence interval not estimable due to insufficient event number greater than Median Value

4. Secondary Outcome: Rate of Complete Response (CRR)
Description: CRR is defined as the percentage of participants who achieve a best response of CR, assessed by IRC per the Lugano Classification
Time Frame: From the date of first dose until end of study (Up to approximately 3 years and 7 months)
Population: Modified safety analysis set
Measure: Median (95% Confidence Interval); unit: Percentage of participants
Groups:
- Tislelizumab: Tislelizumab 200 mg administered IV Q3W until PD unacceptable toxicity, death, or study withdrawal by the participant.
Arm/Group | Tislelizumab
Number analyzed (Participants) | 70
Percentage of participants | 67.1 [54.9 to 77.9]

5. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as the time from the date of the first dose of tislelizumab to the time the response criteria are first met, assessed by IRC per the Lugano Classification
Time Frame: From the date of first dose until end of study (Up to approximately 3 years and 7 months)
Population: Modified safety analysis set; participants with available data were included in the analysis.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Tislelizumab
Number analyzed (Participants) | 61
Weeks | 12.0 [11.86 to 12.29]

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study drug, whether considered related to study drug or not.
  An SAE is any untoward medical occurrence that, at any dose:
  * Results in death.
  * Is life-threatening.
  * Requires hospitalization or prolongation of existing hospitalization
  * Results in disability/incapacity
  * Is a congenital anomaly/birth defect
  * Is considered a significant medical AE by the investigator based on medical judgement
Time Frame: From the date of first dose until end of study (Up to approximately 3 years and 7 months)
Population: The Safety Analysis Set included all participants who received any dose of tislelizumab.
Measure: Number; unit: Participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 70
Participants
  Participants with At least one TEAE | 68
  SAE | 18

7. Secondary Outcome: Number of Participants With Significant Changes in Clinical Laboratory Results
Description: Clinical laboratory (e.g. hematology, serum chemistry, urinalysis) values were evaluated for each laboratory parameter and participants with clinically significant changes are summarized.
Time Frame: From the date of first dose until end of study (Up to approximately 3 years and 7 months)
Population: The Safety Analysis Set included all participants who received any dose of tislelizumab.
Measure: Number; unit: Participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 70
Participants | 0

8. Secondary Outcome: Number of Participants With Significant Changes in Electrocardiograms
Time Frame: From the date of first dose until end of study (Up to approximately 3 years and 7 months)
Population: The Safety Analysis Set included all participants who received any dose of tislelizumab.
Measure: Number; unit: Participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 70
Participants
  Postbaseline corrected QT interval > 450 msec | 0
  ≥ 1 postbaseline electrocardiogram | 21
  Increase corrected QT interval of ≤ 30 msec | 18
  Increase > 30 msec but ≤ 60 msec corrected QT interval | 4

ADVERSE EVENTS:
Time Frame: From the date of first dose until end of study (Up to approximately 3 years and 7 months)
Arm/Group | Tislelizumab
All-Cause Mortality (participants affected / at risk) | 8/70
Serious Adverse Events (participants affected / at risk) | 18/70
Other Adverse Events (participants affected / at risk) | 68/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab (N=70)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (7)
Ascites (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Hepatitis B (Infections and infestations) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Renal injury (Renal and urinary disorders) | 1 (1)
Renal tubular injury (Renal and urinary disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab (N=70)
Anaemia (Blood and lymphatic system disorders) | 9 (18)
Leukopenia (Blood and lymphatic system disorders) | 6 (10)
Lymphopenia (Blood and lymphatic system disorders) | 3 (33)
Neutropenia (Blood and lymphatic system disorders) | 4 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (9)
Hyperthyroidism (Endocrine disorders) | 3 (4)
Hypothyroidism (Endocrine disorders) | 26 (64)
Diarrhoea (Gastrointestinal disorders) | 10 (13)
Nausea (Gastrointestinal disorders) | 6 (7)
Toothache (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 7 (7)
Asthenia (General disorders) | 5 (9)
Chills (General disorders) | 4 (4)
Pyrexia (General disorders) | 40 (55)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (4)
Liver injury (Hepatobiliary disorders) | 3 (7)
Influenza (Infections and infestations) | 4 (7)
Nasopharyngitis (Infections and infestations) | 5 (10)
Pharyngitis (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 27 (72)
Urinary tract infection (Infections and infestations) | 3 (4)
Alanine aminotransferase increased (Investigations) | 14 (34)
Amylase increased (Investigations) | 3 (17)
Aspartate aminotransferase increased (Investigations) | 11 (16)
Bilirubin conjugated increased (Investigations) | 6 (12)
Blood bilirubin increased (Investigations) | 7 (19)
Blood bilirubin unconjugated increased (Investigations) | 5 (14)
Blood creatine phosphokinase increased (Investigations) | 8 (15)
Blood lactate dehydrogenase increased (Investigations) | 4 (4)
Blood thyroid stimulating hormone increased (Investigations) | 8 (11)
Blood uric acid increased (Investigations) | 5 (7)
Gamma-glutamyltransferase increased (Investigations) | 4 (5)
Lymphocyte count decreased (Investigations) | 3 (14)
Neutrophil count decreased (Investigations) | 10 (48)
Neutrophil count increased (Investigations) | 3 (5)
Platelet count decreased (Investigations) | 7 (19)
Weight decreased (Investigations) | 12 (25)
Weight increased (Investigations) | 24 (79)
White blood cell count decreased (Investigations) | 15 (52)
White blood cell count increased (Investigations) | 4 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 (8)
Hyperuricaemia (Metabolism and nutrition disorders) | 10 (21)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (7)
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7)
Headache (Nervous system disorders) | 7 (7)
Hypoaesthesia (Nervous system disorders) | 3 (4)
Paraesthesia (Nervous system disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (20)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (18)
Rash (Skin and subcutaneous tissue disorders) | 11 (15)
Hypertension (Vascular disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT03209973/Prot_001.pdf
  • Statistical Analysis Plan (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT03209973/SAP_000.pdf